CLINICAL TRIAL: NCT01507740
Title: Profile of Soluble and Cellular Biomarkers and of Functional Imaging During Antiangiogenic Therapies in Cancer Patients
Status: Terminated | Type: Observational
Why Stopped: Study was stopped 04.10.2014 prematurly after recruitment of HCC and RCC patients. NSCLC (2 of 10 patients planned) and CRC patients recruitment was stopped
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Wolfgang Hilbe, Prof. Wolfgang Hilbe, Medical University Innsbruck
Other Study IDs: Praemarker AAT 08
Record Dates: First submitted 2009-09-18; First posted 2012-01-11 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Hepatocellular Cancer; Non-small Cell Lung Cancer; Renal Cell Cancer; Colorectal Cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Colorectal Neoplasms | interventions — Bevacizumab; Sorafenib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Consecutive serum and blood probes will be taken and will be examined and correlated with functional imaging and the clinical course. Following parameters have been selected: soluble markers in the plasma (VEGF, bFGF, ICAM, sVGFR-2 IL-8, SDF1 and Dickkopf 3) and cellular parameters like circulating endothelial cells (CEC) and circulating endothelial progenitor cells (CEPs).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Control group n=20
- 2: investigational group (cancer patients) n=40 patients treated with antiangiogenic agent
  Interventions: Drug: Avastin; Drug: Suntent; Drug: Nexavar

INTERVENTIONS:
Drug: Avastin — Dosage, duration, indications and contraindications of treatment rely on the sole responsibility of the treating physician and are not subject of the present study
  Groups: 2
Drug: Suntent — Dosage, duration, indications and contraindications of treatment rely on the sole responsibility of the treating physician and are not subject of the present study
  Groups: 2
Drug: Nexavar — Dosage, duration, indications and contraindications of treatment rely on the sole responsibility of the treating physician and are not subject of the present study
  Groups: 2

SUMMARY:
Tumour angiogenesis has been identified to play a critical role in tumour growth and this knowledge has led to the identification of new targets for cancer therapy. Multiple angiogenic factors are involved in the regulation of angiogenesis, among them VEGF (vascular endothelial growth factor) and its receptor are of crucial relevance. The inhibition of VEGF signaling by monoclonal antibodies or small molecules (kinase inhibitors) has already been successfully established for the treatment of different cancer entities and multiple new drugs are being tested in clinical trials. The ever-expanding list of antiangiogenic agents being available in the near future will raise the questions when to use which agent and in which sequence. As a consequence biomarkers are going to be indispensible tools for choosing the most effective drugs and to predict dosing and resistance.

The present project is based on an academic clinical trial in which patients suffering from different cancer types (colorectal cancer, non-small cell lung cancer, renal cell cancer and hepatocellular cancer) treated routinely with antiangiogenic agents will be included. Consecutive serum and blood probes will be taken and will be examined and correlated with functional imaging and the clinical course. The following parameters have been selected: soluble markers in the plasma (VEGF, bFGF, ICAM, sVGFR-2 IL-8, SDF1 and Dickkopf 3) and cellular parameters like circulating endothelial cells (CEC) and circulating endothelial progenitor cells (CEPs).

In conclusion, the present project is screening for potential biomarkers and biomarker combinations relevant for antiangiogenic drugs in different tumour types. The predictive value of such profiles should then be evaluated in larger cohorts. In the future such profiles could possibly help clinicians to use these agents more effectively and therefore also more economically.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Patients with HCC, NSCLC, RCC or CRC treated with an approved antiangiogenic drug (bevacizumab, sorafenib, sunitinib)*
* Patients with at least one measurable lesion. Lesions must be measurable by CT-scan or MRI (Magnetic resonance imaging) according to Response Evaluation Criteria in Solid Tumours (RECIST)

Exclusion Criteria:

* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must use adequate birth control measures during the course of the trial. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Known or suspected allergy to the investigational agent or any agent given in association with this trial -_> allergy
* MRI contraindications: implants (pacemaker)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * 10 NSCLC patients treated with bevacizumab monotherapy (maintenance therapy)
  * 10 RCC patients treated either with sorafenib or sunitinib monotherapy
  * 10 CRC patients treated with bevacizumab monotherapy
  * 10 HCC patients treated with sorafenib monotherapy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-07; Primary Completion 2012-12 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Progression free survival under antiangiogenic therapy | progression of disease, up to 48 months
  From date of study inclusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Hilbe, Prof, Principal Investigator — Medical University Innsbruck
Locations (1):
- University Hospital Innsbruck, Internal Medicine V, Hematology Oncology, Innsbruck, Austria